CLINICAL TRIAL: NCT04579458
Title: Assessment of COVID (Coronavirus Disease)-19 in Tearfilm
Brief Title: Assessment of COVID-19 in Tearfilm
Status: Withdrawn | Type: Observational
Why Stopped: Not able to enroll the amount required.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Sapna Gangaputra, Assistant Professor of Ophthalmology Co-Fellowship Director Vitreoretinal Diseases and Surgery, Vanderbilt University Medical Center
Other Study IDs: 201127
Record Dates: First submitted 2020-10-06; First posted 2020-10-08 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Covid19; Ophthalmopathy; Eye Diseases
Keywords: Positive COVID 19; Ophthalmology; Eye Diseases
MeSH Terms: conditions — COVID-19; Eye Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 Positive: COVID-19 positive in nasopharyngeal swabs and tears or saliva.
  Interventions: Procedure: Collection of tears and saliva.

INTERVENTIONS:
Procedure: Collection of tears and saliva. — Saliva and ocular tears will be collected.

SUMMARY:
To assess the co-relation of COVID-19 in nasopharyngeal swabs and tears or saliva, and to determine duration of COVID-19 activity in ocular fluid and saliva by serial tests over 3 months.

DETAILED DESCRIPTION:
Patients who underwent COVID-19 testing at VUMC (Vanderbilt University Medical Center) and had provided a written informed consent to be contacted in the future for COVID related studies will be offered participation in this study. The COVID- 19 has low prevalence in ocular fluids (5% of affected patients) but may survive for a long time or replicate in the conjunctiva, even in asymptomatic patients. Patients with viral conjunctivitis are more likely to have COVID-19 RNA (ribonucleic acid) in tears. The use of Schirmer's strips to collect tears for RNA analysis of viruses has been previously validated. VUMC is performing RNA analysis on nasopharyngeal (NP) swabs for COVID-19 at several locations. Several patients (test positive and test negative) have given consent to be contacted for future research purposes and are available in VICTR (Vanderbilt Institute for Clinical and Translational Research) Datamark and Recovery databases. The positive tested patients will receive a Schirmer's strip in the mail at their home to place in both eyes to test eye fluid and receive a tube for saliva while engaging in a zoom session for monitoring of the process.

Methodology: Patients who underwent COVID-19 testing at VUMC and had provided a written informed consent to be contacted in the future for COVID related studies will be offered participation in this study. The first test for eye fluid and saliva will occur at home with remote monitoring. Participants will be mailed a specimen collection kit, engage in a remote session with a study coordinator through a HIPPA (Health Insurance Portability and Accountability Act of 1996)-compliant video meeting and collect specimens under supervision of the study coordinator. Patients will receive a Schirmer's strip to place in both eyes without topical proparacaine, and a tube to collect saliva. The strips are then sent to the lab in universal viral transport media. Patients who have positive COVID-19 RNA in tears will get repeat Schirmer's test every 4 weeks for 3 months- independent of the nasopharyngeal test results. After a 3-month period, they will be offered a clinic visit at VEI (Vanderbilt Eye Institute) for full dilated eye exam, fluorescein angiography and aqueous biopsies. Lab testing for COVID-19 RNA and other ocular inflammatory mediators will be performed by Dr. Johnathan Schmitz's lab at VUMC under standard viral precautions. All lab analysis will be performed under a research protocol and not for clinical assessment or reporting.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent COVID-19 testing at VUMC, tested positive, and had provided a written informed consent to participate in future COVID related studies will be offered participation in this study.

Exclusion Criteria:

* Patients under 18.
* Patients who do not speak Spanish or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent COVID-19 testing at VUMC and tested positive.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
Co-relation of COVID-19 activity | 3 months
  Patients will receive a Schirmer's strip to place in both eyes without topical proparacaine, and a tube to collect saliva. The co-relation of COVID-19 in nasopharyngeal swabs and tears or saliva will be measured and reported by serial tests over 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sapna Gangaputra, Principal Investigator — Vanderbilt Eye Institiute
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Napoli PE, Nioi M, d'Aloja E, Fossarello M. The Ocular Surface and the Coronavirus Disease 2019: Does a Dual 'Ocular Route' Exist? J Clin Med. 2020 Apr 28;9(5):1269. doi: 10.3390/jcm9051269. PMID 32353982
- [Background] Xie HT, Jiang SY, Xu KK, Liu X, Xu B, Wang L, Zhang MC. SARS-CoV-2 in the ocular surface of COVID-19 patients. Eye Vis (Lond). 2020 Apr 26;7:23. doi: 10.1186/s40662-020-00189-0. eCollection 2020. PMID 32355863
- [Background] Khavandi S, Tabibzadeh E, Naderan M, Shoar S. Corona virus disease-19 (COVID-19) presenting as conjunctivitis: atypically high-risk during a pandemic. Cont Lens Anterior Eye. 2020 Jun;43(3):211-212. doi: 10.1016/j.clae.2020.04.010. Epub 2020 Apr 27. No abstract available. PMID 32354654
- [Background] Wu P, Duan F, Luo C, Liu Q, Qu X, Liang L, Wu K. Characteristics of Ocular Findings of Patients With Coronavirus Disease 2019 (COVID-19) in Hubei Province, China. JAMA Ophthalmol. 2020 May 1;138(5):575-578. doi: 10.1001/jamaophthalmol.2020.1291. PMID 32232433
- [Background] Lee SY, Kim MJ, Kim MK, Wee WR. Comparative analysis of polymerase chain reaction assay for herpes simplex virus 1 detection in tear. Korean J Ophthalmol. 2013 Oct;27(5):316-21. doi: 10.3341/kjo.2013.27.5.316. Epub 2013 Sep 10. PMID 24082768
- [Background] WHO. Laboratory testing for 2019 novel coronavirus (2019-nCoV) in suspected human cases - interim guidance. 2020; 2020.
- [Background] Sullivan PS, Sailey C, Guest JL, Guarner J, Kelley C, Siegler AJ, Valentine-Graves M, Gravens L, Del Rio C, Sanchez TH. Detection of SARS-CoV-2 RNA and Antibodies in Diverse Samples: Protocol to Validate the Sufficiency of Provider-Observed, Home-Collected Blood, Saliva, and Oropharyngeal Samples. JMIR Public Health Surveill. 2020 Apr 24;6(2):e19054. doi: 10.2196/19054. PMID 32310815